CLINICAL TRIAL: NCT00569595
Title: Improving Health Habits in Impoverished Populations
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Lillian Gelberg, MD, MSPH, Professor of Family Medicine & Public Health, UCLA Department of Family Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: R21 DK71065 (completed); R21DK071065 (NIH)
Record Dates: First submitted 2007-12-05; First posted 2007-12-07 (Estimated); Last update posted 2011-06-07 (Estimated); Status verified 2011-06

CONDITIONS: Diabetes; Chronic Diseases
Keywords: Prevention of Diabetes and other chronic diseases
MeSH Terms: conditions — Diabetes Mellitus; Chronic Disease | interventions — Counseling

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Multi-Level, Patient-Directed, Lifestyle Change, Health Promotion Program
  Interventions: Behavioral: Self-Care Stimulating Disease Prevention Program
- 2 (Sham Comparator): Patient health counseling program by lay health educators Entitled "Fighting Cancer with Advice."
  Interventions: Behavioral: Fighting Cancer with Advice

INTERVENTIONS:
Behavioral: Self-Care Stimulating Disease Prevention Program — The intervention is aimed at improving diet, increasing physical activity, and reducing sedentary behaviors among low-income patients, assuming that this will increase motivation and self-confidence to adhere to self-care regimens based on personal prioritizing and progressive goal setting.
  Arms: 1
Behavioral: Fighting Cancer with Advice — Patient health counseling program by lay health educators entitled "Fighting Cancer with Advice."
  Arms: 2

SUMMARY:
Poor diet, physical inactivity, and sedentary behaviors among low-income, minority populations have been linked to greater risk of chronic health conditions such as overweight/obesity, cardiovascular disease, and type 2 diabetes. Low-income clinics that serve these populations often represent an untapped opportunity for health promotion in impoverished individuals. This exploratory project proposes to address this scientific gap by introducing and conducting a randomized controlled pilot of the Self-Care Stimulating Disease Prevention Program to address poor dietary habits, physical inactivity, and sedentary lifestyle behaviors among low income, uninsured patient populations.

DETAILED DESCRIPTION:
Poor diet, physical inactivity, and sedentary behaviors among low-income, minority populations have been linked to greater risk of chronic health conditions such as overweight/obesity, cardiovascular disease, and type 2 diabetes. Low-income clinics that serve these populations often represent an untapped opportunity for health promotion in impoverished individuals. Few studies have examined the feasibility of using brief physician advice and multi-level, clinic-based interventions to change poor dietary habits, physical inactivity, and sedentary lifestyle behaviors among these culturally diverse populations that comprise the clinic population. This exploratory project proposes to address this scientific gap by introducing and piloting a Self-Care Stimulating Disease Prevention Program (SCSDPP) to address poor dietary habits, physical inactivity, and sedentary lifestyle behaviors among low income, uninsured patient populations (primarily Latinos) served by the community clinics of the Venice Family Clinic (VFC) health center in Los Angeles County. The program will include the development of 1) a simple-to-use patient Health Priority Assessment (HPA) tool designed to assess patient preferences for behavior change; 2) a standard protocol for physicians to provide brief health advice using motivation interviewing (< 2 minutes per visit); 3) a protocol for distributing self-help aids for patient use (e.g., pedometer, exercise videos); and 4) a series of monthly follow-up counseling sessions by lay health educators (e.g., promotores) to help patients address their lifestyle change priorities over time. We will conduct a randomized controlled pilot of the SCSDPP in approximately 100 patient cases at two community health clinics within the VFC health center system. The pilot will utilize precise outcome measures, including commonly-accepted biomarkers (e.g., HgbA1c, fasting blood glucose) and psychometrically-validated measures of process and health status, to accurately assess the magnitude of changes in diet and physical activity among patients over a 12-month observation period. The feasibility of integrating the SCSDPP into the community health clinic setting will be evaluated, and is the primary aim of this project. The results will inform efforts to plan a larger, successor study. Relevance to Public Health: this study evaluates a clinic-based brief intervention to help prevent overweight/obesity, a public health problem that has been linked to the development of the metabolic syndrome and other precursors of diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18 and older
* English or Spanish-speaking
* Accessible by telephone or in person over time
* Willing to cooperate with data collection
* Planning to be in the Los Angeles area for the next 6 to 12 months so they can complete the study period

Exclusion Criteria:

* Women who are pregnant
* History of cancer, except non-melanoma skin cancer or in situ cancers
* Medical conditions preventing free choice of foods (e.g., colitis, poorly-controlled diabetes)
* Medical conditions precluding participation in common forms of aerobic or resistance exercise (e.g., uncontrolled angina, asthma or hypertension; severe physical impairment; and end-stage disease conditions such as congestive heart failure, nephropathy from any cause, or advanced chronic pulmonary disease)
* Does not show any desire to change any of their health behaviors (i.e., healthy eating, physical activity, sedentary behavior, or control their weight)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2008-11; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Serum glycosylated hemoglobin, heart rate recovery step test | 4 and 6 months

SECONDARY OUTCOMES:
Total Cholesterol, BMI, waist circumference, healthy eating, physical activity, perceived health status, patient satisfaction, mood | 4 and 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Lillian Gelberg, MD, MSPH, Principal Investigator — UCLA Department of Family Medicine
Locations (2):
- United States (2):
  - UCLA Department of Family Medicine, Los Angeles, California
  - Queenscare Family Clinics, Los Angeles, California